CLINICAL TRIAL: NCT01556685
Title: Measuring Neutralizing Antibodies in the Patients Treated With Interferon Beta 1a IM, in Mexico and Colombia
Brief Title: MATRIX: Measuring Neutralizing Antibodies in the Patients Treated With Interferon Beta 1a IM, in Mexico and Colombia
Acronym: MATRIX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: AVX-MEX-09-17
Record Dates: First submitted 2011-10-20; First posted 2012-03-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Avonex (Active Comparator): Approximately 90 subjects treated with IFN beta 1a IM 30μg
  Interventions: Other: clinical and neurological evaluation; Other: Blood Sample; Genetic: Blood Sample
- Group 2 Jumtab (Active Comparator): Approximately 90 subjects treated with IFN beta 1a IM biosimilar
  Interventions: Other: clinical and neurological evaluation; Other: Blood Sample; Genetic: Blood Sample

INTERVENTIONS:
Other: clinical and neurological evaluation — The day of the usual IFN beta 1a IM injection
Other: Blood Sample — For evaluation of interferon-related Nab
Genetic: Blood Sample — genetic evaluation - predisposition to Nab generation

SUMMARY:
This is a cross sectional Phase 4, multicenter, study of AVONEX® and JUMTAB® to determine the frequency of IFN induced Neutralizing Antibodies (Nabs). A secondary component is the long term retrospective observational evaluation conducted to measure efficacy, adherence to therapy, tolerability, and safety in subjects with relapsing MS related to antibody status and treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the frequency of neutralizing antibodies in patients treated with IFN beta 1a IM (Avonex) and IFN beta 1a IM biosimilar formulation (Jumtab).

Secondary objectives:

* Evaluate the effect of Nabs on the severity of the relapses on each treatment group, measured by:

  * The need and duration of steroid courses
  * The need and duration for hospitalization.
* To evaluate the safety and tolerability of the IFN beta 1a IM treatments [Avonex and Jumtab].
* To identify the genetic profile of the patients with relation to the predisposition to Nab development (HLA DR4 (in particular HLADRB1* 0401 and 0408) and DR16 (in particular HLADRB1* 1601)
* At selected sites: To evaluate the influence of the interferon and the Nabs on the activation of neopterin

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for entry into this study, candidates must meet all of the following eligibility criteria at the time of selection:

  * No limitation of age, EDSS or other disease parameters will be applied.
  * Subject with MS
  * Subjects treated with IFN beta 1a IM (Avonex) or the biosimilar formulation of IFN beta 1a IM (Jumtab) in line with the local prescription information
  * The IFN beta 1a IM (Avonex or Jumtab) treatment should be the first disease modifying treatment
  * The subject should be treated with the same drug for at least 18 months and up to a maximum of 3 years

Exclusion Criteria:

* Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of selection:

  * No informed consent
  * Patients with combination therapy (IFN + immunosuppressive therapy)
  * Patients pretreated with immunosuppressive therapy
  * Treatment with any investigational product, including investigational symptomatic therapies for MS (e.g., 4Aminopyridine) and investigational therapies for NonMS indications, during the review period.

NOTE: subjects may receive investigational symptomatic therapies for MS at any time prior to evaluation period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibodies to Interferon beta 1a IM (Avonex) or IFN beta 1a IM biosimilar | Day 1
Percentage of patients with interferon induced Nabs measured in luciferase test | Day 1
neutralizing antibodies to IFN beta 1a IM (Avonex) or IFN beta 1a IM biosimilar formulation (Jumtab) | 1 day
Percent of patients with interferon induced neutralizing antibodies measured in a luciferase test | 1 day

SECONDARY OUTCOMES:
Rate and duration of corticosteroid use for relapse | Day 1
Need and duration of hospitalization for relapse | Day 1
Genetic profile of patients with relation to their predisposition to Nab development | Day 1
The interferon activity will be tested by neopterin protein activation (level before IFNbeta1a IM injection and 48 hours after the injection) | twice measured: - Day 1 before IFN injection - 48-72hours after the IFN injection
Genetic profile of population with relation to predisposition to Nab generation | Day 1
Rate/ duration of corticosteroid use for relapse | measured up to 3 years prior to enrollment @ Day 1
Need/ duration of hospitalization for relapse | measured up to 3 years prior to enrollment @ Day 1
Genetic profile of patients with relation to the predisposition to Nab development | 1 day
Interferon activity will be tested by neopterin protein activation before and after injection | 48-72 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Bogotá, Colombia
- Research Site, León, Guanajuato, Mexico